CLINICAL TRIAL: NCT04415112
Title: Effectiveness of a Mediterranean Diet to Treat Non-Alcoholic Fatty Liver Disease in Children
Brief Title: Mediterranean Diet Treatment for NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2017-234
Record Dates: First submitted 2020-05-27; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Mediterranean Diet
Keywords: Non Alcoholic Fatty Liver Disease; Mediterranean Diet; Low Fat Diet; Children
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Diet, Mediterranean; Diet, Fat-Restricted

STUDY DESIGN:
Intervention Model Description: The study design was a single-blinded randomized, parallel assignment clinical trial of children with NAFLD was conducted. Participants were randomized in a 1:1 fashion to either 12-weeks of a Mediterranean diet or a low fat diet.
Who Masked: Participant
Masking Description: The study design was single blind and the participants did not know what diet they had taken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean Diet (Active Comparator): The MD diet is rich in plant based foods including vegetables, whole cereal and fruit with the main added fat being extra virgin olive oil. In addition, the diet emphasises, while consumption of legumes, nuts and fish is high, consumption of red meat and home-made desserts is low, and consumption of fermented milk and poultry is moderate. The MD diet had a target macronutrient composition of 35-40% fat (with <10% of energy as saturated fat), 40-44% carbohydrate and 20% protein.
  Interventions: Behavioral: Mediterranean Diet
- Low Fat Diet (Active Comparator): The Low Fat diet had a target macronutrient composition of 55% of energy from carbohydrate, 20-25% from fat (with <10% of energy as saturated fat) and 20-25% from protein. Nutrition education focused on choosing foods containing ≤3 grams of fat/serving, limiting added fats, and using low-fat meal preparation strategies. Parents were instructed to offer their children ample amounts of grains, vegetables, fruits, lean meats, low-fat dairy products and limit high-fat foods
  Interventions: Behavioral: Low Fat Diet

INTERVENTIONS:
Behavioral: Mediterranean Diet — A list of foods high consumption of vegetables, fruits, non-refined cereals, legumes and potatoes, moderate consumption of fish and poultry and low consumption of full fat dairies, red meat and its products and homemade sweets.
  Arms: Mediterranean Diet
Behavioral: Low Fat Diet — These children are forbidden to eat high-fat foods such as fried foods, butter, cream cheese, while foods such as fruits, vegetables (starchy and non-starch), cereals, poultry, lean meat and low-fat dairy products are allowed.
  Arms: Low Fat Diet

SUMMARY:
Treatment for Nonalcoholic Fatty Liver Disease (NAFLD) is through lifestyle modification consisting of caloric restriction and exercise, with an emphasis on weight loss. Unfortunately, the success and longevity of lifestyle changes that focus on weight loss, are poor in children. The dietary recommendation of calorie restriction alone may not be optimal in a pediatric population for multiple reasons including changes in hormonal milieu, growth velocity, and decreased bone mineral density that occur with significant weight loss. Mediterranean Diet (MD) is based on the high intake of extra virgin olive oil, vegetables, fruits, cereals, nuts and legumes; moderate intakes of fish and other meats, dairy products and red wine and low intakes of eggs and sweets. So, it provides a large amount of monounsaturated fatty acids, polyunsaturated fatty acids, vegetable proteins, fibre and antioxidants; and low amounts of sugar, cholesterol and saturated fats. It offers a lot of choice in food selection, and well tolerated, and many people can adhere to it over the long term. The investigators aimed to evaluate the effects of a MD vs. low fat diet on changes in hepatic steatosis, aminotransferases, and anthropometric measurements among obese children with NAFLD

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is a disease caused by abnormal lipid accumulation in the liver without alcohol intake or other organic causes. NAFLD covers a range of liver diseases ranging from simple oil infiltration to non-alcoholic steatohepatitis (NASH), fibrosis and cirrhosis. The most important risk factor in the development of NAFLD is insulin resistance due to obesity. Insulin resistance increases hepatic steatosis and accumulation of hepatic fatty acids by increasing peripheral lipolysis and the entry of fatty acids into the liver. In parallel with the increased prevalence of childhood obesity, the occurrence of NAFLD is increasing among children. The risk that the NAFLD can turn into chronic liver disease increases the importance of the disease even more when children become adults Mediterranean Diet (MD) has gained popularity in scientific literature because it is one of the healthiest diets in the world.This diet is based on the high intake of extra virgin olive oil, vegetables, fruits, cereals, nuts and legumes; moderate intakes of fish and other meats, dairy products and red wine and low intakes of eggs and sweets. So, it provides a large amount of monounsaturated fatty acids, polyunsaturated fatty acids, vegetable proteins, fibre and antioxidants; and low amounts of sugar, cholesterol and saturated fats. MD is characterized as low-carbohydrate (40% of calories) and in contrast to low-fat diets, the MD includes fat as 40% of the diet. It offers a lot of choice in food selection, and well tolerated, and many people can adhere to it over the long term. There are a limited number of studies investigating the effectiveness of the MD in NAFLD treatment in different countries. However, there are no studies in the treatment of children with NAFLD in Turkey. The primary aims to this study is to evaluate the effects of a MD vs. low fat diet on changes in hepatic steatosis, aminotransferases, and anthropometric measurements among obese children with NAFLD in Turkey. The secondary aim to this study is to evaluate the effects of the both diets in insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NAFLD
* Body mass index z-score >85th percentile

Exclusion Criteria:

* Secondary causes of NAFLD (eg. medication induced)
* Use of weight loss medications
* Diabetes Mellitus
* Other causes of fatty liver disease (eg. Wilson disease, alpha-1 antitrypsin deficiency, auto-immune hepatitis, and viral hepatitis)

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Non-alcoholic Fatty Liver Disease Ultrasonography Score | 12 weeks
  A semiquantitative score to measure Non-alcoholic Fatty Liver Disease will be used. Degrees of steatosis range from 0 (no steatosis) to 3 (severe steatosis), according to Hamaguchi score, which used a 6-point scoring system based on liver brightness.

SECONDARY OUTCOMES:
Evaluate the effects of the both diets in insulin resistance | 12 weeks
  Changes in Homeostatic Model Assessment of Insulin Resistance from baseline to 12-week post Mediterranean diet and low fat diet intervention
Evaluate the effects of the both diets in capillary blood glucose | 12 weeks
  Changes in fasting capillary blood glucose (mg/dL) from baseline to 12-week post Mediterranean diet and low fat diet intervention
Evaluate the effects of the both diets in fasting insulin levels | 12 weeks
  Changes in fasting insulin (μU/mL) levels from baseline to 12-week post Mediterranean diet and low fat diet intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ulas E Akbulut, Study Chair — Antalya Training and Research Hospital
Locations (1):
- Ulas Emre Akbulut, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Properzi C, O'Sullivan TA, Sherriff JL, Ching HL, Jeffrey GP, Buckley RF, Tibballs J, MacQuillan GC, Garas G, Adams LA. Ad Libitum Mediterranean and Low-Fat Diets Both Significantly Reduce Hepatic Steatosis: A Randomized Controlled Trial. Hepatology. 2018 Nov;68(5):1741-1754. doi: 10.1002/hep.30076. Epub 2018 Oct 14. PMID 29729189